CLINICAL TRIAL: NCT02350101
Title: Introduction of a Massive Transfusion Protocol - Evaluation Over Three Years
Brief Title: Massive Transfusion Protocol With Coagulation Algorithm
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Oliver Theusinger, PD Dr med, University of Zurich
Other Study IDs: KEK-ZH-Nr. 2010-0234/4
Record Dates: First submitted 2015-01-16; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Rotational thromboelastometry — In bleeding patients point of care measurements are performed, in this case Rotational Thromboelastometry (ROTEM) to guide the use of blood products and coagulation factors.

SUMMARY:
In 2008 at the University Hospital Zurich (USZ) a massive transfusion protocol was introduced. Based on laboratory diagnostics and point of care (POC) devices including ROTEM.

Goal of this retrospective study is to evaluate the influence of this algorithm on coagulation, use of blood products, coagulation factors and ROTEM evolution.

DETAILED DESCRIPTION:
In 2008 at the USZ a massive transfusion protocol was introduced. Based on laboratory diagnostics and POC (point of care) devices including ROTEM.

Goal of this retrospective study is to evaluate the influence of this algorithm on coagulation, use of blood products, coagulation factors and ROTEM evolution over three years (2008-2010)

ELIGIBILITY:
Inclusion Criteria:

* Massive transfusion

Exclusion Criteria:

* non

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients needing massive transfusion (more than 10 RBCs)
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Coagulation in ROTEM | 3 years
  Point of care devices are used in bleeding patients. In the university hospital of Zurich an algorithm in the case of massive bleeding was introduced in 2008. The primary outcome measure is to investigate the changes of ROTEM parameters in the sense of amelioration reflected by better coagulation by using goal directed transfusions.

SECONDARY OUTCOMES:
Transfusion needs | 3 years
  To evaluate the blood products and coagulation factors needed and to evaluate if there is a reduction between the time before the introduction of the algorithm compared to afterwards.